CLINICAL TRIAL: NCT05893043
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled Trial of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Multiple Ascending Doses of GSBR-1290 in Japanese and Non-Japanese Healthy Volunteers
Brief Title: A Study of Multiple Ascending Doses of GSBR-1290 in Japanese and Non-Japanese Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gasherbrum Bio, Inc., a wholly owned subsidiary of Structure Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GSBR-1290-03
Record Dates: First submitted 2023-05-30; First posted 2023-06-07 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Study drug (GSBR-1290 or placebo) administration in Cohort 1 is double-blind and Study drug (GSBR-1290) administration in Cohort 2 is open label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: GSBR-1290 or Placebo (Experimental): Healthy Japanese participants will receive once daily doses of study drug (GSBR-1290 or placebo oral capsules) for up to 4 weeks.
  Interventions: Drug: GSBR-1290; Other: Placebo
- Cohort 2: GSBR-1290 (Experimental): Healthy non-Japanese participants (Caucasians or African Americans) will receive once daily doses of study drug (GSBR-1290 oral capsules) for up to 4 weeks.
  Interventions: Drug: GSBR-1290

INTERVENTIONS:
Drug: GSBR-1290 — Participants will receive GSBR-1290 oral capsules.
  Other Names: GSBR-1001290
Other: Placebo — Participants will receive matching placebo oral capsules.
  Arms: Cohort 1: GSBR-1290 or Placebo

SUMMARY:
The purpose of this study is to assess safety and tolerability of multiple oral doses of GSBR-1290 (capsule) in healthy adult Japanese participants compared to non-Japanese participants.

DETAILED DESCRIPTION:
This is a multiple ascending dose (MAD) study in which 4 dose levels will be evaluated in 2 cohorts from Day 1 to Day 28 (4-week period). The starting dose of GSBR-1290 will be based on results from the single ascending dose (SAD) study (GSBR-1290-01) and MAD study (GSBR-1290-02 [NCT05762471]).

ELIGIBILITY:
Inclusion Criteria:

For Cohort 1 only:

1. Japanese participants must have both parents and 4 grandparents of Japanese origin

   For Cohort 2 only:
2. Non-Japanese participants must not have parents and grandparents of Japanese origin. Non-Japanese participants will be limited to Caucasians of European and Latin American descent or African Americans

   For Cohorts 1 and 2:
3. Must have given written informed consent before any study-related activities are carried out
4. Adult males and females, age 18 to 55 years of age (inclusive) at screening
5. Body Mass Index (BMI) greater than or equal to (>=) 18.5 and less than or equal to (<=) 24.9 kilogram per square meter (kg/m^2), with a body weight (to 1 decimal place) >= 45.0 kg at screening
6. No nicotine use
7. Sitting blood pressure after resting for 5 minutes between 90 to 140 millimeter of mercury (mm Hg) systolic and 50 to 90 mm Hg diastolic and a heart rate between 40 to 100 beats per minute
8. Have suitable venous access for blood sampling

Exclusion Criteria:

1. History or presence of significant cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic, or neurological disease, including any acute illness or major surgery within the past 3 months
2. Liver function test results elevated > 2.0-fold the upper limit of normal (ULN) for gamma-glutamyl transferase (GGT), alkaline phosphatase (ALP), aspartate transaminase (AST) or alanine transaminase (ALT). Bilirubin above ULN
3. Estimated glomerular filtration rate (eGFR) < 60 milliliter per minute (mL/min)/1.73m^2 body surface area
4. Known hypersensitivity to any of the study drug ingredients
5. Any other condition or prior therapy that would make the participant unsuitable for this study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2023-04-24 (Actual); Primary Completion 2023-06-28 (Actual); Study Completion 2023-06-28 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs) and Serious AEs | From start of study drug up to End of study (EOS) (up to Day 42)
Number of Participants Based on Severity of AEs | From start of study drug up to EOS (up to Day 42)
Number of Participants With Clinically Significant Change From Baseline in Vital Signs | Baseline up to EOS (Day 42)
Number of Participants With Clinically Significant Change From Baseline in Electrocardiogram (ECG) Parameters | Baseline up to EOS (Day 42)
Number of Participants With Clinically Significant Change From Baseline in Laboratory Parameters | Baseline up to EOS (Day 42)

SECONDARY OUTCOMES:
Analysis of Maximum Observed Plasma Concentration (Cmax) for GSBR-1290 at Specified Timepoints Pre-dose and Post-dose to Calculate Pharmacokinetic (PK) Parameters | 31 days
Analysis of Time to Maximum Observed Plasma Concentration (Tmax) for GSBR-1290 at Specified Timepoints Pre-dose and Post-dose to Calculate PK Parameters | 31 days
Analysis of Plasma Trough Concentrations for GSBR-1290 at Specified Timepoints Pre-dose and Post-dose to Calculate PK Parameters | 31 days
Analysis of Area Under the Plasma Concentration-time Curve (AUC) for GSBR-1290 at Specified Timepoints Pre-dose and Post-dose to Calculate PK Parameters | 31 days

CONTACTS AND LOCATIONS:
Locations (1):
- ACT, Anaheim, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol
Time Frame: Data sharing requests will be considered beginning 36 months after the study publication (manuscript accepted for publication) and either 1) the product have been granted marketing authorization in at least two regulatory jurisdictions, or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Researchers will submit a request containing the research objectives, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). Structure Therapeutics does not grant external requests for individual de-identified patient data for the following purposes:
  * re-evaluating safety and efficacy end points already addressed in the product labelling,
  * assessing safety or efficacy for an indication in current development
  Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a panel of external advisors. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement.